CLINICAL TRIAL: NCT03877796
Title: Development of Drug Response Predictor (DRP) to Test Sensitivity to Investigational Anti-Cancer Drugs in Patients With Advanced Ovarian Cancer
Brief Title: Clinical Pre-screening Protocol for Ovarian Cancer
Status: Recruiting | Type: Observational
Sponsor: Allarity Therapeutics (Industry)
Collaborators: Amarex Clinical Research (Other)
Responsible Party: Sponsor
Other Study IDs: 2X-1000
Record Dates: First submitted 2019-03-14; First posted 2019-03-18 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Samples with archival ovarian cancer tumor tissue is collected for measurement using mRNA or microRNA.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

GROUPS / COHORTS (1):
- Ovarian cancer patients: with formalin-fixed paraffin-embedded (FFPE) tumor tissue available
  Interventions: Device: Drug Response Predictor® (DRP)

INTERVENTIONS:
Device: Drug Response Predictor® (DRP) — A DRP is an assay that based on samples from a tumor can predict whether the tumor will respond to a specific drug or not.

SUMMARY:
The patient's local archival tumor tissue (FFPE) from original tumor, or from the metastatic tissue, will be collected to potentially identify if they - at a later stage of their disease - will be likely to benefit from treatment with any of the investigational cancer drugs available to Allarity Therapeutics. Data from this study can further be used to explore in a retrospective fashion, sensitivity to other chemotherapeutic drugs previously used in the treatment of their ovarian cancer, to investigate whether or not the DRP® method can predict and confirm the obtained sensitivity to the prior given drugs as well as prospective analyses guiding the Investigators on future treatments.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histological confirmed epithelia ovarian cancer
* Patients must have platinum-resistant disease, defined as progression within 6 months after the last dose of platinum-based chemotherapy, or are platinum ineligible.
* Patients have received no more than one prior line of therapy in the platinum resistant or platinum ineligible setting
* FFPE tumor tissue available

Exclusion Criteria:

* Patients who have platinum-refractory disease, defined as progression during the last platinum-based chemotherapy.
* Other malignancy with exception of any stage I and II cancer that is deemed cured by the Investigator

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patients will be identified at their already planned treatment and or at control visits at the oncology department
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2019-04-11 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Identification of ovarian cancer patients with high likelihood of being sensitive to investigational cancer drug | up to 2 years
  based on FFPE ovarian cancer tissue

SECONDARY OUTCOMES:
Retrospective analysis of whether or not the DRP method can predict and confirm the obtained sensitivity to the prior drugs used in the treatment of ovarian cancer | up to 2 years

CONTACTS AND LOCATIONS:
Locations (5):
- United States (3):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - OU Health Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Swedish Center for Research and Innovation, Seattle, Washington
- United Kingdom (2):
  - Beatson West of Scotland Cancer Centre, Glasgow, Scotland
  - Guy's and St Thomas' NHS Foundation Trust, Guy's Hospital, London